CLINICAL TRIAL: NCT05807724
Title: Geriatric Emergency Department Fall Injury Prevention Project
Acronym: GREAT-FALL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida Atlantic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1903012
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Fall; Fall Injury; Emergencies
Keywords: Geriatric
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Current care (No Intervention): Current care at the ED
- Phone-based fall-prevention strategy (Experimental): The phone-based fall-prevention strategy is based on the CDC's Stopping Elderly Accidents Deaths & Injuries (STEADI) program (https://www.cdc.gov/steadi/index.html). The STEADI Algorithm will be the template for both fall-prevention strategies utilized in this study. In addition, the CDC Check For Safety-A Home Prevention Checklist for Older Adults pamphlet will be used.
  At the time of study enrollment, the STEADI program written material will be provided and components of it will be discussed with the study subjects and caregivers, if present.
  The phone-based strategy will provide the patient and caregiver easy to read materials before ED discharge and a structured phone call around 14 days post ED discharge.
  Interventions: Other: Phone-based fall-prevention strategy
- Home-visit fall prevention strategy (Experimental): The specific components of the home-visit fall prevention strategy are similar to the Phone-Based Fall-Prevention Strategy. The essential difference is the in-person visit by the research associate to discuss and reinforce the fall-prevention strategy.
  Interventions: Other: Home-visit fall prevention strategy

INTERVENTIONS:
Other: Phone-based fall-prevention strategy — Written education material and Phone-Based Fall-Prevention Strategy
  Arms: Phone-based fall-prevention strategy
Other: Home-visit fall prevention strategy — Written education material and Home visit-Based Fall-Prevention Strategy
  Arms: Home-visit fall prevention strategy

SUMMARY:
This prospective randomized study will assess an emergency department (ED) based prevention strategy in geriatric patients at high risk for recurrent falls and injury. Falling is a major health hazard in older adults with a number of proposed but unproven protocols to prevent fall-related injuries. This study proposes to study one of these strategies, the CDC's Stopping Elderly Accidents, Deaths and Injuries program (the STEADI Program).

DETAILED DESCRIPTION:
The purpose of this study is to assess whether certain Emergency Department patients at high risk of recurrent falls and injuries related to falls will benefit from the recommendations of the Center for Disease Control and Prevention's (CDC) Stopping Elderly Accidents, Deaths and Injuries program (STEADI Program).

Study subjects will be randomized to one of 3 arms: 1) current care; 2) a phone-based fall-prevention strategy; or 3) a home-visit fall prevention strategy

1. Current emergency department care
2. STEADI recommendations administered via phone at 14 days
3. STEADI recommendations administered via a home visit at 14 days

The STEADI recommendations include the following:

* Follow-up with a primary care physician
* An assessment of your risk of falling. This includes looking at your ability to walk, your strength and balance.
* Assessment medications looking for potential medication interactions
* Measuring your vital signs (blood pressure and heart rate)
* Assessment of your vision
* Assessment of your footwear
* Recommendations to improve home safety (such as ensuring proper lighting, ensuring adequate hand-rails, and others)

Initial data collection will occur at the time of the ED visit. Intervention will occur 14 days after ED visit. Telephonic follow-up will occur at 3 months and 6 months after study enrollment.

Data will be collected from the patients/patient representatives and medical records. All data will be collected by trained research assistants (RAs)

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 65 with a ground level fall who live at home will be eligible for study inclusion

Exclusion Criteria:

* Being transferred from another facility, trauma activation, hospice or palliative care participant, end-stage heart failure (two or more congestive heart failure hospitalizations in past 6 months), end stage emphysema (two or more chronic obstructive pulmonary disease hospitalizations in past 6 months), metastatic cancer, severe leukemia or multiple myeloma or lymphoma on treatment or requiring transfusion and end stage renal disease requiring dialysis. An additional exclusion criterion is patients with dementia, if the subject is unable to state name or unable to point to an object (for those with aphasia)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 644 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Recurrent fall requiring ED revisit at 6 months | 6 months
  Number of Participants with 6 months ED Returns
Fall-related injury at 6 months | 6 months
  Number of Participants with 6 months ED Returns

SECONDARY OUTCOMES:
Specific fall-related injury at 6 months | 6 months
  Number of Participants with 6 months ED Returns
Fall-related mortality | 6 months
  Hospital census data
All-cause mortality | 6 months
  Hospital census data

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Shih, MD, Principal Investigator — Florida Atlantic University
Locations (1):
- Delray Medical Center, Delray Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shankar KN, Liu SW, Ganz DA. Trends and Characteristics of Emergency Department Visits for Fall-Related Injuries in Older Adults, 2003-2010. West J Emerg Med. 2017 Aug;18(5):785-793. doi: 10.5811/westjem.2017.5.33615. Epub 2017 Jul 14. PMID 28874929
- [Background] Bhasin S, Gill TM, Reuben DB, Latham NK, Ganz DA, Greene EJ, Dziura J, Basaria S, Gurwitz JH, Dykes PC, McMahon S, Storer TW, Gazarian P, Miller ME, Travison TG, Esserman D, Carnie MB, Goehring L, Fagan M, Greenspan SL, Alexander N, Wiggins J, Ko F, Siu AL, Volpi E, Wu AW, Rich J, Waring SC, Wallace RB, Casteel C, Resnick NM, Magaziner J, Charpentier P, Lu C, Araujo K, Rajeevan H, Meng C, Allore H, Brawley BF, Eder R, McGloin JM, Skokos EA, Duncan PW, Baker D, Boult C, Correa-de-Araujo R, Peduzzi P; STRIDE Trial Investigators. A Randomized Trial of a Multifactorial Strategy to Prevent Serious Fall Injuries. N Engl J Med. 2020 Jul 9;383(2):129-140. doi: 10.1056/NEJMoa2002183. PMID 32640131
- [Background] Burns E, Kakara R. Deaths from Falls Among Persons Aged >/=65 Years - United States, 2007-2016. MMWR Morb Mortal Wkly Rep. 2018 May 11;67(18):509-514. doi: 10.15585/mmwr.mm6718a1. PMID 29746456
- [Background] Bergen G, Stevens MR, Burns ER. Falls and Fall Injuries Among Adults Aged >/=65 Years - United States, 2014. MMWR Morb Mortal Wkly Rep. 2016 Sep 23;65(37):993-998. doi: 10.15585/mmwr.mm6537a2. PMID 27656914
- [Background] National Prevention Council. Healthy Aging in Action: Advancing the National Prevention Strategy [Internet]. Washington (DC): US Department of Health and Human Services; 2016 Nov. Available from http://www.ncbi.nlm.nih.gov/books/NBK538955/ PMID 30896903
- [Background] Panel on Prevention of Falls in Older Persons, American Geriatrics Society and British Geriatrics Society. Summary of the Updated American Geriatrics Society/British Geriatrics Society clinical practice guideline for prevention of falls in older persons. J Am Geriatr Soc. 2011 Jan;59(1):148-57. doi: 10.1111/j.1532-5415.2010.03234.x. PMID 21226685
- [Background] Crandall M, Duncan T, Mallat A, Greene W, Violano P, Christmas AB, Barraco R. Prevention of fall-related injuries in the elderly: An Eastern Association for the Surgery of Trauma practice management guideline. J Trauma Acute Care Surg. 2016 Jul;81(1):196-206. doi: 10.1097/TA.0000000000001025. PMID 26958795
- [Background] Jung D, Shin S, Kim H. A fall prevention guideline for older adults living in long-term care facilities. Int Nurs Rev. 2014 Dec;61(4):525-33. doi: 10.1111/inr.12131. Epub 2014 Sep 12. PMID 25212122
- [Background] Kruschke C, Butcher HK. Evidence-Based Practice Guideline: Fall Prevention for Older Adults. J Gerontol Nurs. 2017 Nov 1;43(11):15-21. doi: 10.3928/00989134-20171016-01. PMID 29065212
- [Background] Thurman DJ, Stevens JA, Rao JK; Quality Standards Subcommittee of the American Academy of Neurology. Practice parameter: Assessing patients in a neurology practice for risk of falls (an evidence-based review): report of the Quality Standards Subcommittee of the American Academy of Neurology. Neurology. 2008 Feb 5;70(6):473-9. doi: 10.1212/01.wnl.0000299085.18976.20. PMID 18250292
- [Background] Phelan EA, Mahoney JE, Voit JC, Stevens JA. Assessment and management of fall risk in primary care settings. Med Clin North Am. 2015 Mar;99(2):281-93. doi: 10.1016/j.mcna.2014.11.004. PMID 25700584
- [Background] Davenport K, Alazemi M, Sri-On J, Liu S. Missed Opportunities to Diagnose and Intervene in Modifiable Risk Factors for Older Emergency Department Patients Presenting After a Fall. Ann Emerg Med. 2020 Dec;76(6):730-738. doi: 10.1016/j.annemergmed.2020.06.020. Epub 2020 Sep 30. PMID 33010956
- [Background] Cheng P, Tan L, Ning P, Li L, Gao Y, Wu Y, Schwebel DC, Chu H, Yin H, Hu G. Comparative Effectiveness of Published Interventions for Elderly Fall Prevention: A Systematic Review and Network Meta-Analysis. Int J Environ Res Public Health. 2018 Mar 12;15(3):498. doi: 10.3390/ijerph15030498. PMID 29534531
- [Background] Biese KJ, Busby-Whitehead J, Cai J, Stearns SC, Roberts E, Mihas P, Emmett D, Zhou Q, Farmer F, Kizer JS. Telephone Follow-Up for Older Adults Discharged to Home from the Emergency Department: A Pragmatic Randomized Controlled Trial. J Am Geriatr Soc. 2018 Mar;66(3):452-458. doi: 10.1111/jgs.15142. Epub 2017 Dec 22. PMID 29272029
- [Background] Goldberg EM, Marks SJ, Resnik LJ, Long S, Mellott H, Merchant RC. Can an Emergency Department-Initiated Intervention Prevent Subsequent Falls and Health Care Use in Older Adults? A Randomized Controlled Trial. Ann Emerg Med. 2020 Dec;76(6):739-750. doi: 10.1016/j.annemergmed.2020.07.025. Epub 2020 Aug 25. PMID 32854965
- [Background] Ouslander JG, Reyes B, Diaz S, Engstrom G. Thirty-Day Hospital Readmissions in a Care Transitions Program for High-Risk Older Adults. J Am Geriatr Soc. 2020 Jun;68(6):1307-1312. doi: 10.1111/jgs.16314. Epub 2020 Jan 29. PMID 31994723